CLINICAL TRIAL: NCT03649009
Title: Thiamine As An Adjuvant Therapy For Hyperlactatemia In Septic Shock Patients: A Prospective Randomized Study
Brief Title: Thiamine As An Adjuvant Therapy For Hyperlactatemia In Septic Shock Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universiti Kebangsaan Malaysia Medical Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FF-2017-389
Record Dates: First submitted 2018-07-05; First posted 2018-08-28 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Hyperlactatemia
Keywords: Thiamine; Lactate; Septic shock
MeSH Terms: conditions — Hyperlactatemia; Shock, Septic | interventions — Saline Solution; Thiamine; Hydrocortisone; Adrenal Cortex Hormones; Metoclopramide

STUDY DESIGN:
Intervention Model Description: This study is a prospective, randomized controlled trial
Who Masked: Participant
Masking Description: This study is a single-blinded trial, with the participants from both intervention and placebo group will be masked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Normal Saline (Placebo Comparator): Normal Saline 50 mls infused over 1 hour 3 times per day for total 3 days for placebo group after recruitment and randomization done.
  If patients develop rashes or redness after normal saline administration, IV hydrocortisone (corticosteroid) 200mg stat dose will be given.
  Interventions: Other: Normal Saline; Drug: Hydrocortisone
- IV Thiamine (Active Comparator): IV Thiamine 200mg diluted in 50mls normal saline infused over 1 hour 3 times per day for total 3 days for Thiamine group after recruitment and randomization done.
  If patients develop nausea after thiamine administration, IV metoclopramide (antiemetic)10mg stat dose will be given. If patients develop redness and rashes after Normal Saline infusion, IV hydrocortisone (corticosteroid) 200mg stat dose will be given.
  Interventions: Drug: Thiamine; Drug: Hydrocortisone; Other: Metoclopramide

INTERVENTIONS:
Other: Normal Saline — Normal Saline 50 mls infused over 1 hour 3 times per day for total 3 days after recruitment and randomization.
  Arms: Normal Saline
Drug: Thiamine — IV Thiamine 200 mg diluted in 50 mls normal saline infused over 1 hour 3 times per day for total 3 days after recruitment and randomization
  Other Names: Vitamin B1
  Arms: IV Thiamine
Drug: Hydrocortisone — If patient develop redness or rashes after normal saline infusion, IV hydrocortisone 200 mg stat will be given
  Other Names: Corticosteroid
Other: Metoclopramide — If patient develop nausea after IV thiamine infusion, IV metoclopramide 10mg stat will be given. If patient develop redness or rashes after normal saline infusion, IV hydrocortisone 200 mg stat will be given.
  Other Names: Maxolon
  Arms: IV Thiamine

SUMMARY:
The study aimed to assess the effectiveness of intravenous thiamine as compared with placebo in reducing the lactate level in septic shock patients.

DETAILED DESCRIPTION:
Introduction

Thiamine (Vitamin B1) is an essential component for cellular metabolism. It circulates in our body as free thiamine as well as active phosphorylated form - thiamine pyrophosphate (TPP). TPP acts as a co-factor for mitochondrial oxidative decarboxylation process and glycolytic pathway. In the deficient/ absence of thiamine, anaerobic metabolism occurs and causing lactate production with severe biochemical derangement.

Thiamine deficiency has shown to be more prevalent in critically ill patients, with rates ranging from 20 % to 70 % . The deficient might due to the lack of intake or increased losses. Patients who had previous bariatric surgery or gastrointestinal disorders such as peptic ulcer disease, Crohn's disease and bowel obstruction will suffer from thiamine deficiency due to malabsorption. In addition, malnutrition related to oncology, prolonged parenteral nutrition without adequate vitamin supplementation, septic shock patients with renal replacement therapy In septic shock, there is often associated with macro and micro-circulatory dysfunctions causing tissue hypoperfusion with elevation of serum lactate. A study done by Puskarich et al (2013) showed that early lactate normalization (within 6 hours) was an independent predictor of survival in patients treated for sepsis and septic shock. Nguyen et al (2004) also showed that early lactate clearance within 12 hours of resuscitation had twofold reduction of the relative risk of death for severe sepsis patients. Therefore, Surviving Sepsis Guidelines in 2016 had included early lactate clearance within first 6 hours of resuscitation will be the goal of treatment resuscitation.

A study done by Donnino et al (2010) concluded that there was an association of low thiamine levels with lactic acidosis in septic shock patients. In general, the lactate level of 2.0-2.5 mmol/L is considered elevated, however when the lactate level raised > 4mmol/L it is considered 'high' with corresponding lactic acidosis (pH < 7.35). With lactic acidosis, severe cardiovascular adverse effects of hemodynamic instability, myocardial depression and reduced responsiveness to the inotropic supports and vasopressors will occured.

In view of the severity of lactic acidosis with thiamine deficiency, Donnino et al in 2016 studied intravenous thiamine as the resuscitation drug for septic shock patients and found that there was significantly reduced lactate at 24 hours for patients with thiamine deficiency. However, there were no significant differences in the lactate level in patients with normal baseline of thiamine level.

According to the European Society for Clinical Nutrition and Metabolism (ESPEN) guideline for parenteral nutrition in intensive care, all patients who suspected of thiamine deficiency were recommended to receive thiamine supplementation of 100 to 300 mg/day during the first 3 days in the ICU. A literature review by Dinicolantonio et al (2013) also suggested that thiamine supplementation up to 200 mg three times a day in cases of proven deficiency among heart failure patients. In addition, European Federation of Neurological Societies (EFNS) recommended that in particular for Wernicke encephalopathy patients, intravenous thiamine dose of up to 600mg/day (200 mg three times daily) was recommended without significant adverse events reported.

In view of the importance of normalizing the serum lactate, and the current lacking evidence of thiamine in sepsis management, therefore we aimed to use the higher effective dose in order to achieve a good reduction of serum lactate level as well as to improve overall patient's outcome in septic shock.

Methodology

All septic shock patients that admitted to GICU, UKKMC during the study period will be screened for possible enrollment based on the inclusion and exclusion criteria. For the eligible patients, written informed consent will be obtained from the patient itself or from his/her legal guardian.

Following enrollment, the recruited patients will be randomly assigned into 2 groups, thiamine group (TG) or a placebo group (PG) by using computer-generated randomization program. Arterial and central venous catheterization will be performed as a routine, with haemodynamic support continued in both groups following the Surviving Sepsis Campaign (SSC) protocol 2016 for sepsis and septic shock patients. Thiamine group (TG) will be receiving intravenous thiamine 200 mg diluted in 50 ml of normal saline whereas placebo group will receive 50 ml of normal saline only. It will be infused over 1 hour and administered 3 times/day for total 3 days duration. If patient developed nausea after thiamine adminstration, IV metoclopramide 10mg stat will be given. However, if patient developed rashes or redness after normal saline administration, IV hydrocortisone 200mg stat will be given. The study drug will be commenced after recruitment and randomization done.

Arterial blood sample will be collected in a heparinised blood-gas syringe by trained ICU staff nurse at enrolment (time 0) before commencing study drug, 12 hours and 24 hours thereafter. A blood sample will then be analyzed immediately by using a blood gas analyzer in ICU (ABL 800 Basic, Radiometer Medical ApS, Denmark). Following that, other blood parameter includes full blood count, renal function and coagulation-related variables and clinical variables required for determination of the APACHE II score and SOFA score will be documented. Subsequent serum lactate level will be recorded for 3 consecutive days.

Primary outcomes are to assess the relative lactate level change from baseline to 24 hours after the initiation of the study medication dose (defined as (lactate at 0 hour-lactate at 24 hours)/lactate at 0 hour x100%) and to assess the rate of lactate change over 24 hours. Additional outcomes included time to shock reversal (time for weaning off all vasopressors), APACHE II score at 0 and 24 hours and SOFA score at 3 consecutives days, ICU length of stay and in hospital mortality. Any use of renal replacement therapy/ dialysis will also be examined.

Statistical analysis

Sample size calculation The sample size was calculated by using power and sample size calculation (PS) software program based on reduction of lactate level in 24 hours between placebo and thiamine treatment group in a previous study by Donnino et al (2016) Requested output: Sample size Design: Independent Alpha = 0.05, power= 80% δ =1, ợ = 2.2, m = 1 Case sample size for each group = 30 Total sample size: 30 x 2 plus 20% drop-out rate = 72

Therefore, this study will require 36 treatment subjects and 36 control subjects be able to reject the null hypothesis with probably (power) 0.8. Type I error probability associated with this test of this null hypothesis is 0.05.

Statistical tests All statistical data will be performed using IBM SPSS for Windows, version 24.0 (IBM Corp, rmonk, N. Y,USA). Continuous data will be analyzed using independent T-test or Mann-Whitney U test as appropriate. Chi square test will be used to analyze categorical data. Mixed model ANOVA analysis will be performed to determine the effect of treatment of thiamine in reduction of lactate level over 24 hours and the difference of means between group variables. A value of p<0.05 will be considered as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old
2. Septic shock patients 16 (Definition: Sepsis( presence of two or more q Sequential Organ Failure Assessment with documented/suspected infection) and hypotension requiring use of vasopressors to maintain MAP≥ 65 mmHg and having serum lactate ≥ 2 mmol/L despite adequate fluid resuscitation (> 30mls/kg of crystalloid within the first 3 hours)

Exclusion Criteria:

1. Patients with a known allergy to the study drug.
2. Pregnant patients
3. Patients with limitation of therapy
4. Patients with liver failure (include acute liver failure described as development of coagulopathy, international normalized ratio ( INR) of greater than 1.5, any degree of mental alteration( encephalopathy) in a patient without preexisting cirrhosis and with an illness of less than 26 weeks duration 17 or class C Child Pugh classification with the score of 10-15.18 )

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-12-01 (Estimated); Study Completion 2019-03-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of the relative lactate level change over 24 hours | 0 -24 hours during the study drug administration
  To assess the relative lactate level change from baseline to 24 hours after the initiation of the study drugs (defined as (lactate at 0 hour-lactate at 24 hours)/lactate at 0 hour x100%).
  Arterial blood sample for lactate will be collected in a heparinised blood-gas syringe by trained ICU staff nurse at enrolment (time 0) before commencing study drug, and 24 hours after the study drug administration. A blood lactate sample will be analyzed by using a blood gas analyzer in ICU (ABL 800 Basic, Radiometer Medical ApS, Denmark).

SECONDARY OUTCOMES:
Assessment of the time for shock reversal | From the date of randomization until the date of first documented weaning off the inotropes or date of death from any cause, whichever came first, assessed up to 100 weeks
  Assessment of the duration used for weaning off the vasopressors in hours. It will be calculated from the date and time of the inotropes started until the date and time of the inotropes stopped
Assessment of the disease severity | 0- 24 hours after recruitment and randomization
  To assess APACHE (Acute physiology and Chronic Health Evaluation) II score to predict the patient mortality. APACHE II score consists of 12 variables with maximum score of 72. The higher the score, the higher the risk of patient's mortality.
Assessment of patients' length of stay | From the date of randomization until the date of either discharged from ICU or death from any cause, whichever came first, assessed up to 100 weeks.
  After patient was recruited, patient will be assessed the total length of stay in ICU in terms of days
Assessment of the disease severity | 0 - 72 hours after recruitment and randomization
  To assess SOFA (sequential organ failure assessment) score to predict patient's mortality risk. The higher the score, the higher the mortality risk.
  SOFA score is based of the degree of 6 organ dysfunction with maximum score of 24.
  Assessment will recorded from the time 0 (after recruitment and randomization) and at 24 hours, 48 hours, and 72 hours.
Assessment of the rate of the lactate change over 72 hours | 0-72 hours during the study drug administration
  To assess the rate of the lactate change over 72 hours after study drug administration.

CONTACTS AND LOCATIONS:
Overall Officials: Cheah SK DR, M. D., Principal Investigator — Universiti Kenangsaan Malaysia Medical Centre
Locations (1):
- Universiti Kebangsaan Malaysia Medical Centre, Cheras, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Starting from 3 month after publication
Access Criteria: Share the information once approval from the publisher